CLINICAL TRIAL: NCT05301920
Title: A Single-center, Open-label, Clinical Effect Observational Study to Evaluate the Safety and Effectiveness of Reducing the Frequency of Migraine Onset Through Clinical Application of Elexir (Trigeminal Nerve Electrical Stimulator) in Migraine Patients
Brief Title: The Evaluation of the Transcutaneous Electrical Stimulation Medical Device's Safety and Effectiveness in Treating the Patients With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nu Eyne Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NE_MIG_001
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): N=20 60Hz pulse electrical stimulation The clinical trial device performs a personal electrical stimulation around the trigeminal nerves for 4weeks (6 times/week), 20 minutes each time.
  Interventions: Device: Elexir (trigeminal nerve electrical stimulator)

INTERVENTIONS:
Device: Elexir (trigeminal nerve electrical stimulator) — Elexir performs a personal electrical stimulation around the trigeminal nerves for 4weeks (6 times/week), 20 minutes each time.

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of trigeminal nerve electrical stimulator on reducing the frequency of migraine onset. It is applied to migraine patients and analyzes the results by comparing them before and after 4weeks.

DETAILED DESCRIPTION:
* Duration of study period (per participant): Screening period (-6~0weeks), Intervention period (4weeks).
* Patient needs to visit site at least 3 times (Screening, Baseline, V4), V2 can be done with screening visit. V3 is tele-Visit.
* The clinical trial device performs a personal electrical stimulation around the trigeminal nerves for 4weeks (6 times/week), 20 minutes each time.
* During the study period, examination and treatment methods are carried out in the same way.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 19 years old
* Patients with migraine with or without migraine aura who meet ICHD-III (2018) diagnostic criteria 1.1 1.2
* Patients with history of migraine more than 1 year
* Patients who have headaches at least twice a month
* Those who do not take migraine prevention drugs from 12 weeks before screening to the end of the study, or who can maintain migraine prevention drugs during clinical trials without changing or adding additional migraine prevention drugs
* A person who voluntarily agreed to participate in this clinical trial

Exclusion Criteria:

* Those who are diagnosed with primary headaches (exception: low-frequency intermittent tension type headaches) and secondary headaches in addition to migraine headaches
* Those who are diagnosed with medication overuse headache in addition to migraine headaches
* Pregnant or lactating of women within 6months
* Among female subjects who are likely to be pregnant, those who disagree to contraception in a medically permitted manner during this clinical trial period. *Medically permitted contraception: condom, Oral contraception that lasted for at least 3 months, contraceptive injection, contraceptive implant, intrauterine device, etc
* Patients with mental illness who can interfere with their participation in the study.
* In the case where medical devices for clinical trials cannot be applied due to being sensitive to orbital nerve stimulation.
* Patients with a history of drug or alcohol abuse
* Those who participated in other clinical trials within 30 days of screening.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Change in the number of days of moderate to severe headache | baseline, 4 weeks
  Check the number of days of moderate to severe headache at 4 weeks after start compared to baseline

SECONDARY OUTCOMES:
Change in the number of headache days | baseline, 4 weeks
  Check the number of headache days in 4 weeks after the start of stimulation compared to the baseline
Change in the frequency of headache days | baseline, 4 weeks
  Check the frequency of headache days in 4 weeks after the start of stimulation compared to the baseline
Change in the frequency of taking the acute phase drug | baseline, 4 weeks
  Check the frequency of taking the acute phase drug in 4 weeks after the start of stimulation compared to the baseline
Change in pain intensity when headache occurs | baseline, 4 weeks
  Check the change in pain intensity when headache occurs in 4 weeks after the start of stimulation compared to the baseline
Change in the headache effect assessment (HIT-6) score | baseline, 4 weeks
  Check the change in the headache effect assessment (HIT-6) in 4 weeks after the start of stimulation compared to the baseline
Change in the migraine-related quality of life (MSQ 2.1) score | baseline, 4 weeks
  Check the migraine-related quality of life (MSQ 2.1) change in 4 weeks after the start of stimulation compared to the baseline
  MSQ 2.1 measures the impact of migraine across three essential aspects. The MSQ total and scale score varies between 0 and 100 with higher scores indicating higher impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No